CLINICAL TRIAL: NCT05984550
Title: The Exploratory Study on the Nicotinamide Mononucleotide (Vital NAD ) to Promote the Rejuvenation of the Peripheral Blood Immune Cells of Adults.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Collaborators: Shanghai Mengchao Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH2301-A-02
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Enhance Immune Function
Keywords: NMN; NAD+; NADH
MeSH Terms: interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated group (Experimental): NMN(Vital NAD) treated group
  Interventions: Drug: NMN

INTERVENTIONS:
Drug: NMN — NMN (Nicotinamide Mononucleotide) is a naturally occurring bioactive nucleotide with the full name of Nicotinamide mononucleotide. Its structure can be divided into α and β Two isomers, of which only β- NMN is a naturally occurring form with biological activity.
  In human body, NMN is the precursor of NAD+(Nicotinamide adenine dinucleotide, also known as coenzyme I), and its function is mainly reflected through NAD+.
  Other Names: Nicotinamide mononucleotide

SUMMARY:
The purpose of this study is to investigate the changes in adult peripheral blood immune cell subpopulations, subpopulations, and cell functional status before and after intervention with Nicotinamide Mononucleotide (Vital NAD ) as NAD+ supplement for a certain period of time。To Explore and validate the biological functions of Nicotinamide Mononucleotide (Vital NAD ) of rejuvenation of the Peripheral blood immune cells of Adults.

DETAILED DESCRIPTION:
This study focuses on the effects of Nicotinamide mononucleotide (Vital NAD) as NAD+ supplement on the subtypes and biological functions of immune cells of Adults, especially the types and subsets of immune cells, immune cell differentiation, and immune cell status indicators. Therefore, this study plans to enroll approximately 20 adult subjects in a daily dose of 600mg/day and receive 30 days of Nicotinamide Mononucleotide (Vital NAD) intervention. The study will evaluate the improvement effect of NMN intervention on human immune cell research indicators before and after intervention. The study will also study the impact of NMN on Hematology and blood biochemical indicators, and evaluate the changes of human Hematology biological age after NMN intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male/females of 18 to 80 years of age.
2. Able to provide written Informed Consent.
3. BMI 25.0-44.9 kg/m².
4. Able to follow verbal and written study directions.
5. Must not be taking or be willing to take any supplements containing any form of niacin for seven days prior to baseline and for the duration of the study.
6. Able to maintain consistent diet and lifestyle habits according to the study.

Exclusion Criteria:

* 1. Diabetes.

  2.Premenopausal or menopause <1 year.

  3.Persons who have received hormone replacement therapy within the past 6 months.

  4.Persons who take vitamin B supplementation and are not willing to discontinue supplementation for 3 weeks before and during the entire study period.

  5.Unstable weight (>3% change during the last 2 months before entering the study).

  6.Significant organ system dysfunction or disease.

  7.Present cancer or history of cancer that has been in remission for <5 years.

  8.Polycystic ovary syndrome.

  9.Major psychiatric illness.

  10.Use of medications known to affect study outcome measures (e.g., steroid) or increase the risk of study procedures (e.g., anticoagulants) that cannot be temporarily discontinued for the study.

  11.Metal implants.

  12.Persons who consume >14 units of alcohol per week.

  13.Unable or unwilling to follow the study protocol or who, for any reason, is considered an inappropriate candidate for the study by the research team.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Nicotinamide mononucleotide (Vital NAD) in whole blood. | before and after at least 30 days of treatment of Vital NAD
Changes in NAD+ and NADH concentrations in whole blood. | before and after at least 30 days of treatment of Vital NAD]
The change of Blood cell indicators TBNK cells of the healthy adults at the points before and after intervention. | before and after at least 30 days of treatment of Vital NAD
The change of Blood biochemical indicators of the healthy adults at the points before and after intervention. | before and after at least 30 days of treatment of Vital NAD
The change of Peripheral blood immune T cells phenotype of the healthy adults at baseline. | before and after at least 30 days of treatment of Vital NAD
The change of Tnaïve, Tscm, Tcm and Tem in peripheral blood of the healthy adults at the points before and after intervention. | before and after at least 30 days of treatment of Vital NAD
The change of SITR1 expression in immune cells of peripheral blood at the points before and after intervention. | before and after at least 30 days of treatment of Vital NAD

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR